CLINICAL TRIAL: NCT07113392
Title: A Multicenter, Randomized, Double-Blind, Active-Controlled Clinical Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Suraxavir Marboxil for Suspension in Pediatric Patients (2 to <12 Years) With Uncomplicated Influenza
Brief Title: A Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Suraxavir Marboxil for Suspension
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangxi Kvvit Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GP681-S-202501
Record Dates: First submitted 2025-07-23; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suraxavir Marboxil (Experimental): Participants will receive a single oral dose of Suraxavir Marboxil on Day 1 based on body weight.
  Interventions: Drug: Suraxavir Marboxil
- Oseltamivir (Active Comparator): Participants will receive oseltamivir twice a day for 5 days based on body weight.
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Suraxavir Marboxil — Suraxavir Marboxil will be administered as oral suspension: 40 mg (if weight ≥ 32 kg), or 20 mg (if weight <32 kg).
  Arms: Suraxavir Marboxil
Drug: Oseltamivir — Oseltamivir will be administered as oral granules: 30 mg (if weight ≤15 kg), 45 mg (if weight > 15 kg to ≤ 23 kg), 60 mg (if weight > 23 kg to ≤ 40 kg) or 75 mg (if weight > 40 kg), twice daily (BID) for 5 days.
  Arms: Oseltamivir

SUMMARY:
This study will evaluate the safety, efficacy and pharmacokinetics of Suraxavir Marboxil compared with oseltamivir in Pediatric Patients (2 to <12 Years) with Uncomplicated Influenza.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged 2 to 12 years (≥2 years and <12 years).
2. body weight≥10 kg at screening.
3. Diagnosed with influenza virus infection based on the following criteria:

   * Positive rapid antigen test (RAT) result from a throat or nasal swab for influenza virus (rapid nucleic acid tests or other rapid molecular diagnostic tests are also acceptable); and
   * Fever at screening (tympanic temperature ≥38.0°C or axillary temperature ≥37.5°C). If antipyretics were taken, fever must be present >1 hour after administration, or If fever subsided (tympanic <38.0°C or axillary <37.5°C) after antipyretic use, fever must have recurred >4 hours after administration; and
   * Presence of at least one moderate or more severe respiratory symptom at screening (including cough, and/or nasal congestion or rhinorrhea).
4. Time interval between the onset of illness symptoms and enrollment is ≤48 hours.

   Onset of illness: defined as the time of the first temperature increase (tympanic temperature ≥38.0°C or axillary temperature ≥37.5°C) or time of first appearance (or caregiver observation) of at least one respiratory symptom associated with influenza virus infection.
5. The participant's legal guardian agrees to the child's participation in the clinical study and signs the informed consent form (ICF). Participants aged ≥8 years must also voluntarily sign the ICF.
6. The investigator assesses that the participant and/or the caregiver can comply with the protocol requirements, follow-up visits, and complete all study procedures and evaluations (e.g., completing the diary card).

Exclusion Criteria:

1. Known hypersensitivity to the active ingredient or excipients of the investigational product.
2. Patients diagnosed with severe or critical influenza at screening: (1) Severe influenza cases were defined by the presence of one or more of the following conditions: a. Dyspnea and/or tachypnea without fever: >30 breaths/min (age >5 years), >40 breaths/min (age 2-5 years).b. Altered mental status (e.g., lethargy, agitation, seizures).c. Severe vomiting/diarrhea with moderate-to-severe dehydration.d. Concurrent pneumonia.e. Significant exacerbation of pre-existing comorbidities.(2) Critical influenza cases were defined by the presence of one or more of the following conditions: a. Respiratory failure.b. Acute necrotizing encephalopathy.c. Septic shock.d. Multiorgan dysfunction.e. Other life-threatening conditions requiring intensive care.

   Note: Based on "Expert Consensus on Diagnosis and Treatment of Influenza in Children (2020 Edition)".
3. History of gastrointestinal diseases affecting drug absorption (e.g., reflux esophagitis, chronic diarrhea, inflammatory bowel disease, intestinal tuberculosis, gastrinoma, short bowel syndrome, post-gastrectomy).
4. Bronchitis, pleural effusion, or interstitial pneumonia suspected by investigator or confirmed by chest imaging.
5. Use of anti-influenza antiviral drugs within two weeks before screening (e.g., neuraminidase inhibitors [oseltamivir, zanamivir, peramivir], cap-dependent endonuclease inhibitors [baloxavir marboxil], hemagglutinin inhibitors [arbidol], M2 inhibitors [amantadine, rimantadine], or other NMPA-approved anti-influenza agents).
6. Clinically relevant abnormal results in physical examination, 12-lead ECG, vital signs, hematology, clinical biochemistry, or urinalysis at screening, which in the investigator's judgment may pose a risk to the participant's safety, affect the study results, or impact the participant's ability to complete the study.
7. Acute respiratory infection (excluding current influenza), otitis media, or sinusitis within 2 weeks pre-screening.
8. Co-infection requiring systemic antibiotics or other systemic therapy at screening.
9. Known/suspected active primary/secondary immunodeficiency (including HIV infection, hematologic malignancies causing severe immunodeficiency).
10. Known or suspected congenital abnormalities of the heart or lungs, or severe primary diseases affecting the cardiovascular, hepatic, renal, or hematopoietic systems, or evidence of active liver disease, including but not limited to jaundice or AST/ALT levels exceeding two times the upper limit of normal (ULN) at screening.
11. Positive serology for hepatitis B surface antigen or a history of hepatitis B infection at screening.

    (Note: participants with HBV vaccination history and no prior HBV infection are exempt from this exclusion after medical history review).
12. History of mental illness, intellectual disability, substance abuse, or other adverse conditions (e.g., inability to read, understand, or write) that, in the investigator's judgment, may limit participation in the study.
13. Influenza vaccination within 6 months pre-screening or planned during the study. (Note: Vaccination history must be verified by medical history review).
14. Participation in any interventional clinical trial (drug/device) within 30 days pre-screening.
15. Intolerance to skin puncture, fainting at the sight of blood or needles, or poor venous access for blood collection at screening.
16. Any other condition deemed unsuitable by the investigator.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | up to Day 15
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Time to Alleviation of Symptoms (TTAS) | up to Day 15
  Defined as the time from treatment initiation until meeting all criteria below for ≥21.5 consecutive hours:
  1. Return to afebrile status (tympanic temperature ≤37.2°C);
  2. Absence/Mild severity for all respiratory symptoms (cough, nasal congestion, rhinorrhea) on the Canadian Acute Respiratory Illness and Flu Scale (CARIFS);
  3. "Yes" response to: "Has your child resumed normal daily activities as before illness?" in the Daily Activity Questionnaire.
Time to Viral Clearance | up to Day 6
  Time from treatment initiation until first undetectable viral titer (below the lower limit of quantification, LLOQ).
Viral Clearance Rate | Days 2, 3,6
  Proportion of participants with viral titers below LLOQ at D2, D3 (if applicable), and D6 (if applicable).
Proportion of patients with influenza viral RNA positivity (by Q-PCR) and measurable viral titers at each time point(D2, D3 if applicable, D6 if applicable). | Days 2, 3,6
  The percentage of patients positive for virus RNA by Q-PCR. Virus titer was quantified from nasopharyngeal swabs by tissue culture methods.
Area Under the Concentration (AUC) of virus RNA by Q-PCR and AUC of virus titer | Up to Day 6
  AUC of the viral load by Q-PCR and AUC of viral titer measured from baseline to Day 6
Change From Baseline in Virus RNA (Q-PCR) at Each Time Point | Days 2, 3,6
  Nasopharyngeal swabs were obtained for viral quantitation.
Time to return to normal activities of daily life | Up to Day15
  Defined as the time between the initiation of the study treatment and the return to normal activities of daily life.
Time to Resolution of Individual Symptoms | Up to Day15
  Time until absence/mild severity (CARIFS 16-item scale) for individual symptoms, sustained ≥21.5h.
Time to Resumption of Normal Daily Activities | Up to Day15
  Time until "Yes" response to the Daily Activity Questionnaire.
Incidence of Influenza-Related Complications | Up to Day15
  Including hospitalization, death, sinusitis, bronchitis, otitis media, and radiologically confirmed pneumonia.
Palatability Assessment of Suraxavir Marboxil using Visual Analog Scale (VAS) | Day1
  Acceptability of taste assessed by 100-mm Visual Analog Scale (VAS) where 0 = "Very bad", 20 = "Bad", 50 = "Neutral", 80 = "Good", 100 = "Very good". Outcome reported as proportion of subjects with VAS score ≥50 (acceptable threshold) .
Grittiness Assessment of Suraxavir Marboxil using Visual Analog Scale (VAS) | Day1
  Perception of grittiness (grainy texture) assessed by 100-mm Visual Analog Scale (VAS) where 0 = "Severe grittiness", 20 = "Grittiness", 50 = "Slight grittiness", 80 = "No grittiness", 100 = "Smooth texture". Outcome reported as proportion of subjects with VAS score ≥50 (acceptable threshold) .
Pharmacokinetic (PK) Endpoints | Up to Day6
  Plasma concentrations of Suraxavir Marboxil and its primary metabolite Suraxavir

IPD SHARING:
Plan to Share IPD: No